CLINICAL TRIAL: NCT03438136
Title: Adult Broad Learning Experiment (ABLE): Feasibility Study
Acronym: ABLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Riverside (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Rachel Wu, Assistant Professor, University of California, Riverside
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1320181
Record Dates: First submitted 2018-01-28; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Half of the participants will participate in the intervention, and the other half will be assigned to a no contact control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): This arm will be enrolled in the intervention.
  Interventions: Behavioral: Adult Broad Learning Experiment (ABLE)
- No intervention arm (No Intervention): This arm will be enrolled in a no contact control group.

INTERVENTIONS:
Behavioral: Adult Broad Learning Experiment (ABLE) — This intervention implements six factors from early childhood experiences: individualized scaffolding (having a responsive teacher), forgiving environment (allowing the learner to make and learn from mistakes), growth mindset (believing that abilities can develop with effort), open-minded learning (exploring new experiences), serious commitment to learning (adopting a "learning" lifestyle), and learning multiple skills simultaneously.
  Arms: Intervention arm

SUMMARY:
This study evaluates the feasibility of enrolling and retaining older adults in a 15-week intervention that will implement six factors from early childhood experiences: individualized scaffolding (having a responsive teacher), forgiving environment (allowing the learner to make and learn from mistakes), growth mindset (believing that abilities can develop with effort), open-minded learning (exploring new experiences), serious commitment to learning (adopting a "learning" lifestyle), and learning multiple skills simultaneously. These six factors will be implemented via concurrent classes at the UCR Extension center (OSHER Lifelong Learning Institute).

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Fluent in English
* Have not been diagnosed with a cognitive condition (e.g., Mild Cognitive Impairment, Alzheimer's, and Dementia)
* Currently not experiencing a mental health disorder (e.g., anxiety, depression, Schizophrenia)
* Have normal eye vision or corrected-to-normal eye vision
* Not proficient in any of the three skills that will be taught during the intervention. Proficiency of skills will be determined by participants' self-report of their experience with each skill. Only potential participants who self-report having less than one or more years of experience with any of the three skills in the past 10 years or as having less than 5 years of experience more than 50 years ago will be considered as being "unfamiliar" with that skill (or skills) and will be qualified to participate in the study.

Exclusion Criteria: n/a

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-12-13 (Estimated); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
Screening-to-enrollment ratio | Beginning of the intervention (Week 1)
  Number of participants we screen relative to the number of participants who enroll
Intervention adherence | Throughout the intervention (15 weeks)
  Amount of homework hours logged and class attendance
Enjoyment of intervention activities | Week 15
  Assessed via a brief questionnaire of 4 questions created by our research team. Range: 4-24, summed across 4 questions.

SECONDARY OUTCOMES:
Executive Function | Pre-test to post-test (15 weeks: Week 1; Week 15)
  Measured by NIH EXAMINER battery
Broad Learning Adult Questionnaire | Pre-test to post-test (15 weeks: Week 1; Week 15)
  New questionnaire developed by PI

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Riverside, Riverside, California, United States